CLINICAL TRIAL: NCT05600699
Title: Long-term Efficacy and Safety Research of Left Bundle Branch Pacing
Status: Completed | Type: Observational
Sponsor: Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Xinhua Li, Deputy director of Cardiology, Linyi People's Hospital
Other Study IDs: Linyi People's Hospital
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Atrioventricular Block; Left Bundle Branch Pacing
MeSH Terms: conditions — Atrioventricular Block | interventions — Pacemaker, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- left bundle branch potential group: the left bundle branch potential was recorded at implantation
  Interventions: Device: Cardiac pacemaker and Select Secure lead
- Purkinje potential group: the purkinje potential was recorded at implantation
  Interventions: Device: Cardiac pacemaker and Select Secure lead
- no-potential group: no potential was recorded at implantation
  Interventions: Device: Cardiac pacemaker and Select Secure lead

INTERVENTIONS:
Device: Cardiac pacemaker and Select Secure lead — model 3830, 69cm, Medtronic, Inc., Minneapolis, MN, USA

SUMMARY:
Patients with successful left bundle branch pacing in our center were included in this study from April 2018 to December 2019. Baseline data was collected, and pacing parameters, ECG and echocardiographic results were analyzed during 3 years follow-up. According to whether or not a potential was recorded and the specific potential characteristics at implantation, the patients were divided into 3 groups: left bundle branch potential group; Purkinje potential group; and no-potential group. During the 3 years follow-up, the investigators collected the ECG、UCG and pacemaker parameters to analyze.

DETAILED DESCRIPTION:
A total of 136 patients with a high percentage of ventricular pacing and successful left bundle branch pacing were included in this study from April 2018 to December 2019. Baseline data was collected, and pacing parameters, ECG and echocardiographic results were analyzed during 3 years follow-up. According to whether or not a potential was recorded and the specific potential characteristics at implantation, the patients were divided into 3 groups: left bundle branch potential group (L group) 31.6%; Purkinje potential group (P group) 10.3%; and no-potential group (N group) 58.1%. During the 3 years follow-up, the investigators collected the ECG、UCG and pacemaker parameters to analyze.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were predicted to require a high percentage of ventricular pacing in our center were enrolled in this study

Exclusion Criteria:

* Low rate of pacing, and loss to follow-up

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From April 2018 to Dec 2019, consecutive patients who were predicted to require a high percentage of ventricular pacing in our center were enrolled in this study. Main indications for the enrolment of patients are atrioventricular block and heart failure (HF) combined with complete left bundle branch block (LBBB). All patients were accorded with indications for pacing therapy of 2013 European Society of Cardiology guidelines on cardiac pacing. The study conforms to the guiding principles of the Declaration of Helsinki and was approved by Ethics Committee of the Linyi People's Hospital. All patients signed the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in left atrium diameter at 3 years | Baseline and 3 years
  Echocardiography is measured by a professional using an ultrasound machine, record the following results: left atrium diameter (ms)
Change from Baseline in left ventricular end diastolic diameter at 3 years | Baseline and 3 years
  Left ventricular end diastolic diameter (ms)
Change from Baseline in left ventricular ejection fraction at 3 years | Baseline and 3 years
  Left ventricular ejection fraction (%)
Change from Baseline in pulmonary artery systolic pressure at 3 years | Baseline and 3 years
  Pulmonary artery systolic pressure (mmHg)

SECONDARY OUTCOMES:
Change from Baseline in threshold at 3 years | Baseline and 3 years
  Threshold was measured with a pace-sensing analyser: threshold (V) at 0.5ms
Change from Baseline in impedance at 3 years | Baseline and 3 years
  Impedance was measured with a pace-sensing analyser: impedance(Ω)

CONTACTS AND LOCATIONS:
Overall Officials: Fingming Li, Study Chair — Linyi People's Hospital
Locations (1):
- Linyi People's Hospital, Linyi, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
all collected IPD would be shared after publishing

REFERENCES:
- [Background] Huang W, Chen X, Su L, Wu S, Xia X, Vijayaraman P. A beginner's guide to permanent left bundle branch pacing. Heart Rhythm. 2019 Dec;16(12):1791-1796. doi: 10.1016/j.hrthm.2019.06.016. Epub 2019 Jun 22. No abstract available. PMID 31233818
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. A Novel Pacing Strategy With Low and Stable Output: Pacing the Left Bundle Branch Immediately Beyond the Conduction Block. Can J Cardiol. 2017 Dec;33(12):1736.e1-1736.e3. doi: 10.1016/j.cjca.2017.09.013. Epub 2017 Sep 22. PMID 29173611
- [Background] Su L, Wang S, Wu S, Xu L, Huang Z, Chen X, Zheng R, Jiang L, Ellenbogen KA, Whinnett ZI, Huang W. Long-Term Safety and Feasibility of Left Bundle Branch Pacing in a Large Single-Center Study. Circ Arrhythm Electrophysiol. 2021 Feb;14(2):e009261. doi: 10.1161/CIRCEP.120.009261. Epub 2021 Jan 9. PMID 33426907
- [Background] Hou X, Qian Z, Wang Y, Qiu Y, Chen X, Jiang H, Jiang Z, Wu H, Zhao Z, Zhou W, Zou J. Feasibility and cardiac synchrony of permanent left bundle branch pacing through the interventricular septum. Europace. 2019 Nov 1;21(11):1694-1702. doi: 10.1093/europace/euz188. PMID 31322651
- [Background] Ponnusamy SS, Muthu G, Kumar M, Bopanna D, Anand V, Kumar S. Mid-term feasibility, safety and outcomes of left bundle branch pacing-single center experience. J Interv Card Electrophysiol. 2021 Mar;60(2):337-346. doi: 10.1007/s10840-020-00807-w. Epub 2020 Jul 4. PMID 32623624